CLINICAL TRIAL: NCT01058694
Title: Adherence to ARV Treatment and Its Effects on Medium Run Socio-Economic Outcomes: Evidence From Western Kenya
Brief Title: The Impact of Short Message Services (SMS) on ARV Adherence in Western Kenya
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Moi Univeristy (Other); World Bank (Other); Indiana University (Other); Harvard University (Other); Columbia University (Other); University of California, San Diego (Other); University of North Carolina (Other)
Responsible Party: James Habyarimana, PhD/Assistant Professor, Georgetown Public Policy Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-005
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: AIDS; Antiretroviral Therapy; Medication Adherence; HIV Infections
Keywords: Mobile phones,; Medication Adherence; Micro-Electrical-Mechanical Systems; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Weekly SMS, brief message (Experimental): Weekly SMS received on Monday at 12 noon
  Interventions: Behavioral: Short Message Services to Support ARV therapy adherence
- Control Group (Active Comparator): Receives a phone, but no messages.
  Interventions: Behavioral: Short Message Services to Support ARV therapy adherence
- Daily SMS, Brief message (Experimental): Receive daily brief message at 12 noon: "This is your reminder"
  Interventions: Behavioral: Short Message Services to Support ARV therapy adherence
- Daily SMS, Long Message (Experimental): Receive a daily long message at 12 noon: "This is your reminder + encouragement"
  Interventions: Behavioral: Short Message Services to Support ARV therapy adherence
- Weekly SMS, Long Message (Experimental): Weekly message sent at 12 noon on Mondays: "This is your reminder + encouragement"
  Interventions: Behavioral: Short Message Services to Support ARV therapy adherence

INTERVENTIONS:
Behavioral: Short Message Services to Support ARV therapy adherence — Short message services were sent to randomly selected consenting subjects on ARV therapy. The frequency and content of the message is varied in a factorial design.

SUMMARY:
The purpose of proposed research is to implement a randomized study that will allow us to understand and address a number of key barriers to patient adherence as well as study the effects of better adherence on health and socio-economic outcomes.

DETAILED DESCRIPTION:
Several studies have shown that proper adherence to treatment regimens is essential for the effectiveness of ARV therapy (e.g Wools-Kaloustian et al. 2006). There is also evidence in that in some treatment programs in Africa, adherence rates are not always high (Gill et al. 2005). Even in settings where adherence levels are found to be high, numerous factors have been identified as being relevant, although the causal effects are unknown (Castro, 2006). As ARV treatment programs are scaled up in Africa, it is essential to understand the socio-economic determinants of adherence to ARV treatment, as well as the impact of interventions to support high levels of adherence. A secondary objective of this study is to understand the socio-economic impacts of higher adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been on ARV therapy at the Chulaimbo Rural Health Center for a maximum of three months and providing consent to participate in the study.

Exclusion Criteria:

* Patients who had been on ARV therapy for more than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
MEMS Adherence | 12 months follow up

SECONDARY OUTCOMES:
Frequency/incidence of ARV treatment interruptions | 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: John Sidle, MD, Principal Investigator — Indiana University; Duncan Ngare, Phd, Principal Investigator — Moi University; Harsha Thirumurthy, Phd, Principal Investigator — University of North Carolina; Markus Goldstein, Phd, Principal Investigator — World Bank; Joshua Graff-Zivin, Phd, Principal Investigator — University of California, San Diego; Damien de Walque, Phd, Principal Investigator — World Bank; Cristian Pop-Eleches, Phd, Principal Investigator — Columbia University; David Bangsberg, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Chulaimbo Rural Health Center, Kisumu, Maseno District, Kenya

REFERENCES:
- [Derived] Pop-Eleches C, Thirumurthy H, Habyarimana JP, Zivin JG, Goldstein MP, de Walque D, MacKeen L, Haberer J, Kimaiyo S, Sidle J, Ngare D, Bangsberg DR. Mobile phone technologies improve adherence to antiretroviral treatment in a resource-limited setting: a randomized controlled trial of text message reminders. AIDS. 2011 Mar 27;25(6):825-34. doi: 10.1097/QAD.0b013e32834380c1. PMID 21252632